CLINICAL TRIAL: NCT04897009
Title: Evaluating the Impact of Neoadjuvant Chemotherapy on the Peripheral Blood Immune Phenotype in Patients With Operable Breast Cancer (ENHANCE)
Brief Title: Impact of Neoadjuvant Chemotherapy on the Peripheral Blood Immune Phenotype in Operable Breast Cancer
Acronym: ENHANCE
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MC200302; NCI-2021-04162 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA116201 (NIH); 20-010563 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Invasive Breast Carcinoma
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Basic science (biospecimen collection): Patients undergo blood sample collection at baseline (prior to first NAC treatment), after taxane and prior to first dose of A/C (for patients receiving a taxane), end of NAC, 1-4 weeks and 6 months post-surgery. Patients also undergo tissue collection at 1-4 weeks and 6 months post-surgery.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and tissue collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This early phase I trial evaluates the impact of chemotherapy before surgery (neoadjuvant) on the peripheral blood immune phenotype in patients with operable breast cancer. Collecting blood and information from patients with breast cancer may help to understand how the immune system influences response to treatment, and how the immune system reacts to breast cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether pre-neoadjuvant chemotherapy (NAC) peripheral blood immune phenotypes (defined by mass cytometry) are associated with pathologic complete response (pCR) after neoadjuvant chemotherapy in patients with operable breast cancer.

II. To evaluate whether the baseline peripheral blood immune phenotype differs between patients with breast cancer and age-matched healthy controls.

SECONDARY OBJECTIVES:

I. To characterize changes in the baseline peripheral blood immune phenotype that arise as a consequence of neoadjuvant chemotherapy.

II. To create a biorepository of peripheral blood samples for future research in breast cancer, including circulating tumor deoxyribonucleic acid (ctDNA), epigenetic and functional studies.

EXPLORATORY OBJECTIVE:

I. To evaluate differences in peripheral blood immune phenotype of patients with oligometastatic breast cancer compared to patients with stage I-III breast cancer.

OUTLINE:

Patients undergo blood sample collection at baseline (prior to first NAC treatment), after taxane and prior to first dose of anthracycline/cyclophosphamide (A/C) (for patients receiving a taxane), end of NAC, 1-4 weeks and 6 months post-surgery. Patients also undergo tissue collection at 1-4 weeks and 6 months post-surgery.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically confirmed, operable, invasive breast cancer. Note: Patients with oligometastatic breast cancer (up to 3 isolated distant metastases) will be eligible after review and approval by principal investigator (PI)
* Recommended to receive neoadjuvant systemic treatment by their primary medical oncologist and planning to receive one of the regimens
* Provide written informed consent
* Willing to return to Mayo Clinic for breast cancer surgery
* Willingness to provide mandatory blood specimens for future research on breast cancer at Mayo Clinic

Exclusion Criteria:

* Patients who have already initiated neoadjuvant chemotherapy for the current malignancy
* Inability to provide blood samples based on the judgement of the treating physician
* Inability to comply with the protocol
* Patient is pregnant or plans to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed, operable, invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Association of peripheral blood immune phenotypes with pathological complete response | Up to 5 years
  For each of the ten unique family subtypes, and individual cell population within a histological subtype, will utilize a logistic regression model to identify those markers measured at baseline that are predictive of achieving a pathological complete response. Will also perform classification and regression trees (CART) modeling to get at the interplay of the markers (i.e. cell subtypes), which are all uniformly expressed as percentages.
Difference of peripheral blood immune phenotypes | Up to 5 years
  Will be assessed between patients with breast cancer and age-matched healthy controls. Will compare the average difference in the baseline marker expression between the cases and age-matched healthy controls using a two-sample t-test. The two-sample t-test will be used to test the null hypothesis of no difference in means against the alternative hypothesis that there is a difference in means; the two-sided P-value will be reported. Will also perform CART modeling as in the first co-primary objective to get at the interplay of the markers.

SECONDARY OUTCOMES:
Changes in baseline peripheral blood immune phenotype as a consequence of neoadjuvant chemotherapy (NAC) | Baseline up to 2-4 weeks post-surgery
  Will calculate the absolute change for each of the 30 markers, including grouped by the ten unique family subsets. In this largely descriptive analysis, within each histologic subtype, the expression levels will be graphically displayed over time (e.g. plotting the median at each of the three occasions, as well as plotting the mean change from baseline at post-NAC and post-surgery; the patient-level trajectories will be superimposed. Because this is a hypothesis generating objective, all data will be graphed and tabulated and any inferential statistics calculated will be limited and should be interpreted with caution.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto A. Leon-Ferre, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials